CLINICAL TRIAL: NCT07006753
Title: Transvaginal Diverticulum Wall Filling and Coverage Technique for Treating Female Circumferential Urethral Diverticulum
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, De-yi Luo, Prof, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025692
Record Dates: First submitted 2025-05-22; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Circumferential Female Urethral Diverticulum
Keywords: circumferential female urethral diverticulum; Transvaginal surgery; Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transvaginal Diverticulum Wall Filling and Coverage Technique (Experimental): Transvaginal Diverticulum Wall Filling and Coverage Technique for Circumferential UD
  Interventions: Procedure: Transvaginal Diverticulum Wall Filling and Coverage Technique

INTERVENTIONS:
Procedure: Transvaginal Diverticulum Wall Filling and Coverage Technique — This surgical intervention is a modified transvaginal technique for the treatment of circumferential female urethral diverticulum (UD). Instead of performing a complete diverticulectomy, the procedure utilizes the patient's own demucosalized diverticular wall to fill the diverticular cavity and reinforce closure of the ostium. The technique aims to preserve the integrity of the dorsal urethra, reduce the risk of fistula, minimize dead space, and improve functional outcomes such as continence and sexual function. This approach is specifically designed for circumferential UD, which poses unique anatomical and surgical challenges.

SUMMARY:
The goal of this clinical study is to learn if a new surgical technique called transvaginal diverticular wall filling and covering is effective and safe for treating circumferential urethral diverticulum (UD) in female patients. The main questions it aims to answer are:

Does this technique reduce the risk of postoperative complications, such as fistula formation or stress urinary incontinence (SUI)? Does it improve urinary symptoms and sexual function? What are the recurrence rates after surgery using this approach?

Researchers will follow two groups of patients:

One group includes patients who had this surgery in the past 5 years (retrospective group).

The other group includes patients who are newly treated with this technique and followed prospectively.

Participants will:

Undergo the transvaginal wall filling and covering surgery. Have regular follow-up visits to assess symptoms, complications, and quality of life.

Complete questionnaires about urinary and sexual function.

DETAILED DESCRIPTION:
Circumferential UD is a rare and complex subtype that surrounds the urethra and is associated with a higher risk of surgical complications when treated with conventional diverticulectomy. To address these challenges, this study utilizes a modified surgical approach in which the demucosalized diverticular wall is preserved, folded, and used to obliterate the diverticular cavity and reinforce the closure of the ostium. This technique aims to reduce surgical trauma, preserve urethral function, minimize dead space, and improve postoperative urinary and sexual function.

All enrolled patients will undergo this standardized surgical intervention. Follow-up assessments will be conducted at predefined timepoints (1 month and 6 months postoperatively). Evaluations will include physical examinations, symptom assessments, and validated questionnaires addressing urinary symptoms, sexual function, and overall quality of life.

Primary and secondary outcome measures include:

Improvement or resolution of UD-related symptoms (e.g., dysuria, dyspareunia, urgency) Incidence of postoperative complications (e.g., urethrovaginal fistula, de novo stress urinary incontinence) Clinical and imaging-confirmed recurrence Patient-reported outcomes regarding urinary and sexual function

This study aims to provide clinical evidence on the feasibility, safety, and potential advantages of this novel technique for managing circumferential urethral diverticulum in women.

ELIGIBILITY:
Inclusion Criteria:

Female patients with imaging-confirmed circumferential urethral diverticulum (UD).

Availability of complete medical records. Minimum of 6 months postoperative follow-up.

Exclusion Criteria:

Presence of uterine prolapse. Diagnosis of vaginitis. Presence of vaginal tumors. Abnormal coagulation function.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Global Response Assessment (GRA) | 6 months postoperatively
  Overall subjective improvement will also be documented using a 5-point Global Response Assessment (GRA) scale:
  1. = Markedly worse
  2. = Slightly worse
  3. = No change
  4. = Slightly improved
  5. = Markedly improved
Recurrence Rate of Urethral Diverticulum Assessed by Clinical Symptoms | 6 months postoperatively
  Recurrence will be assessed within 6 months postoperatively based on:
  Return of typical urethral diverticulum (UD) symptoms, such as:
  Post-void dribbling Dyspareunia Dysuria Recurrent urinary tract infections Palpable anterior vaginal wall mass
Urinary Continence Status Assessed by Symptom Type and Stress Test | 6 months postoperatively
  Urinary continence status will be evaluated at 6 months postoperatively based on:
  Patient-reported urinary symptoms, including the presence or absence of:
  Stress urinary incontinence (SUI): involuntary leakage of urine during physical effort, sneezing, or coughing
  Urgency urinary incontinence (UUI): involuntary leakage accompanied by or immediately preceded by urgency
  Objective cough stress test performed in the lithotomy position with a comfortably full bladder
  Patients will be classified into one of the following categories:
  Continent: No symptoms of SUI or UUI and negative stress test
  SUI: Symptomatic stress incontinence or positive stress test
  UUI: Symptoms consistent with urgency-related leakage
  Mixed urinary incontinence: Presence of both SUI and UUI symptoms

SECONDARY OUTCOMES:
Complications | 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Deyi Luo, PhD, Study Chair — West China Hospital
Locations (1):
- Sichuan University West China Hospital Department of Urology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided